CLINICAL TRIAL: NCT05160623
Title: Treatment of Blepharitis With Povidone-Iodine 1% : a Randomized Controlled Trial
Brief Title: Treatment of Blepharitis With Povidone-Iodine 1%
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Elishai Assayag, Principal investigator, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18004714
Record Dates: First submitted 2021-11-30; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Anterior Blepharitis
MeSH Terms: interventions — Povidone-Iodine; Solutions

STUDY DESIGN:
Intervention Model Description: A prospective, controlled, randomized, observer-masked study. One eye will be allocated for the studied treatment, and the fellow (control) eye will receive the standard treatment.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study eyes (Experimental): Once-daily eyelid hygiene with povidone-iodine 1%
  Interventions: Drug: Povidone-Iodine 1 % Topical Solution
- Control eyes (Active Comparator): Once-daily eyelid hygiene with available lid wipes
  Interventions: Drug: Eyelid cleansing wipes

INTERVENTIONS:
Drug: Povidone-Iodine 1 % Topical Solution — Povidone-Iodine 1 % topical solution on a makeup remover pad, used to clean the lids and lashes once daily
  Arms: Study eyes
Drug: Eyelid cleansing wipes — EYECARE FORTE eyelid wipes (Dr. Fischer, Israel), used to clean the lids and lashes once daily
  Arms: Control eyes

SUMMARY:
One hundred blepharitis patients will be recruited. Each patient will treat one eye once daily with 1% PVI for 30 days by scrubbing the eyelid margin with the solution. The fellow eye will serve as the control and be given the standard treatment (commercial eye wipes). Before treatment initiation, various ocular surface variables will be assessed, such as dry eye grading, subjective discomfort scales, ocular surface questionnaire, and other clinical signs. After 30 days, an identical evaluation will be performed.

DETAILED DESCRIPTION:
Blepharitis is a chronic and very common inflammation of the eyelid margin affecting patients of all ages. This condition can be categorized anatomically (anterior- skin and eyelashes, posterior- meibomian glands), and pathophysiologically (staphylococcal, seborrheic, parasitic [Demodex mites], and meibomian gland dysfunction [MGD]). Combined forms of the disease are not uncommon. Signs and symptoms include itching, redness, flaking, and crusting of the lids, along with ocular surface disturbances such as irritation, dryness, tearing, and corneal damage.

Since no definitive cure is available, treatment recommendations for blepharitis focus on management. They may include eyelid hygiene using warm compresses and scrubbing, topical corticosteroids, topical and oral antibiotics, and dietary adjustments.

Povidone-iodine (PVI) is a widely used antimicrobial agent. Utilization of PVI is prevalent in disinfection of the eye and surrounding skin before intraocular procedures such as cataract surgeries and intravitreal injections. The antiseptic properties of PVI enable it to effectively reduce ocular surface and conjunctival colonization of various pathogens. Therefore, novel uses of ocular PVI seem promising, and some were already assessed in clinical studies.

The optimal concentration of PVI is also a matter of debate. High concentration solutions (5-10%) have greater potency, yet they increase corneal endothelial and epithelial toxicity. Although they may require repeated applications, low concentration solutions (0.1-1%) were proven to be safer and effective and are widely utilized in some countries. However, data regarding the option of treating blepharitis with PVI are lacking, as no comparative or controlled studies have been published to date.

In this study, the aim is to investigate the efficacy of lid scrubbing with PVI 1% in the treatment of anterior blepharitis

This is a prospective, controlled, randomized, observer-masked study. The allocated eye will be specified in a sealed envelope, given to the patient upon recruitment to the study. All investigators will be masked to the treated eye for the duration of the study. The fellow eye will serve as the control. Before treatment initiation, all outcomes will be assessed (specified below). Eligible participants will be assigned to use 1% PVI once daily on either the right or left eye for 30 days. During the first week of treatment, patients will be called to ensure the correct eye is being treated. Patients will be instructed to clean the eyelids and lashes of the study eye with 1% PVI using makeup remover pads (will be supplied to patients). Following treatment, patients will remove residual PVI with a wet makeup pad. The fellow eye (control eye) will receive regular treatment for blepharitis: eyelashes cleansing with commercially available eyelid wipes. Patients will be invited to a follow-up examination after 30 days. All outcomes will be re-assessed after 30 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Anterior or mixed (anterior + posterior) blepharitis.
* Similar clinical condition of both eyes.

Exclusion Criteria:

* Any ocular surface disease other than blepharitis.
* Known allergy to iodine.
* Eye surgery in the last 6 months.
* Ocular trauma in the last 6 months.
* Use of contact lenses in the last 6 months.
* Pregnancy or lactation.
* Daily use of makeup on lashes.
* Any ocular or systemic medication that might affect the ocular microbiota (antibiotics, immunosuppressants, steroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Blepharitis signs on slit-lamp examination | Day 0 (recruitment)
  0-4 grading of each sign (normal, mild, moderate, severe, very severe): eyelid edema, eyelid erythema, scaling and crusting, meibomian glands clogging.
Blepharitis signs on slit-lamp examination | Day 30 (follow-up)
  0-4 grading of each sign (normal, mild, moderate, severe, very severe): eyelid edema, eyelid erythema, scaling and crusting, meibomian glands clogging.

SECONDARY OUTCOMES:
OSDI score | Day 0 (recruitment)
  0-100 score based on the ocular surface disease index (OSDI) questionnaire
OSDI score | Day 30 (follow-up)
  0-100 score based on the ocular surface disease index (OSDI) questionnaire
Subjective eye complaints | Day 0 (recruitment)
  visual analog scale (VAS, 0-10 cm) of subjective eye complaints: itching, dryness, overall discomfort.
Subjective eye complaints | Day 30 (follow-up)
  visual analog scale (VAS, 0-10 cm) of subjective eye complaints: itching, dryness, overall discomfort.
TBUT | Day 0 (recruitment)
  tear break-up time on slit-lamp examination (TBUT, 0-10 seconds)
TBUT | Day 30 (follow-up)
  tear break-up time on slit-lamp examination (TBUT, 0-10 seconds)
National Eye Institute/Industry (NEI) grading scale | Day 0 (recruitment)
  corneal staining- according to NEI grading system (0-15 score, 0-normal. 15-worse)
National Eye Institute/Industry (NEI) grading scale | Day 30 (follow-up)
  corneal staining- according to NEI grading system (0-15 score, 0-normal. 15-worse)
Schirmer's test | Day 0 (recruitment)
  with topical anesthetic (5 minutes, >10mm is normal)
Schirmer's test | Day 30 (follow-up)
  with topical anesthetic (5 minutes, >10mm is normal)

CONTACTS AND LOCATIONS:
Overall Officials: Elishai Assayag, MD, Principal Investigator — Department of Ophthalmology, Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Ophthalmology clinic, Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No